CLINICAL TRIAL: NCT02010762
Title: The Effect of Vitamin D3 to Maintain Surgical Remission in Postoperative Crohn's Disease: a Placebo-controlled Randomized Trial
Brief Title: The Effect of Vitamin D3 to Maintain Surgical Remission in Postoperative Crohn's Disease
Acronym: DETECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Geert D'Haens, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL.45391.018.13
Record Dates: First submitted 2013-12-10; First posted 2013-12-13 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Vitamin D; Postoperative; Recurrence; Inflammatory bowel disease; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Colonic Diseases; Intestinal Diseases; Pathologic Processes
MeSH Terms: conditions — Crohn Disease; Recurrence; Inflammatory Bowel Diseases; Gastroenteritis; Gastrointestinal Diseases; Digestive System Diseases; Colonic Diseases; Intestinal Diseases; Pathologic Processes | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator): Weekly Vitamin D3 drops 25.000 IU for 6 months following ileocoecal resection
  Interventions: Drug: Vitamin D
- Placebo (Placebo Comparator): Weekly placebo drops for 6 months following ileocoecal resection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — 25.000 IU oral drops
  Arms: Vitamin D
Drug: Placebo — placebo oral drops
  Arms: Placebo

SUMMARY:
The majority of patients with Crohn's disease (CD) need to undergo surgical bowel resection. Postoperative recurrence of the disease is virtually inevitable and continues to be one of the most challenging therapeutic problems in inflammatory bowel diseases. Medical treatments to prevent recurrence have had limited effect. Anti-tumor necrosis factor (TNF) agents appear promising but are hampered by immunogenicity, side effects and high cost.

Vitamin D has recently received a lot of scientific attention and was found to have strong anti-inflammatory and antifibrotic effects in gut and liver inflammation. Many CD patients appear to have deficiency in Vitamin D. A controlled trial to prevent relapse of CD in medical (not surgical) remission suggested a preventive effect for Vitamin D but marginally missed its endpoint because of lack of power.

The ultimate proof of the anti-inflammatory effect of Vitamin D in CD can best be studied in the prevention of postoperative recurrence.

DETAILED DESCRIPTION:
Our objective is to study the prophylactic effect of Vitamin D3 to prevent post-operative recurrence of Crohn's disease (CD), with an endoscopic endpoint 6 months after surgery as the primary outcome. Endoscopy has been an established surrogate marker for future clinical relapse. Secondary objectives include clinical recurrence rates at 6 months, the difference in recurrence rates among patients with and without low Vitamin D levels at baseline, the effects of Vitamin D3 on quality of life parameters, resource use and related costs.

ANTICIPATED OUTCOME This study will provide proof of the anti-inflammatory effect of vitamin D, which to our opinion can best be studied in a post-operative setting. Since post-operative recurrence is frequent, a safe and cost-effective therapy is highly needed for this indication. The hypothesis is that patients who receive vitamin D treatment will have less frequent and less severe endoscopic recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years, either male or female
* Established CD
* First or second ileocolonic resection with ileocolonic anastomosis and removal of all tissue macroscopically affected by CD according to the surgeon
* Able to give written informed consent
* Normal levels of serum calcium at inclusion
* Being able to resume oral intake within 2 weeks after surgery

Exclusion Criteria:

* Patients in whom not all visible CD has been resected
* Active fistulizing perianal disease (requiring anti TNF treatment)
* Extensive small bowel resection
* Third, fourth or later ileocolonic resection
* Patients undergoing ileocoecal resection in the Lir!c Trial (NTR 1150, http://www.trialregister.nl/trialreg/admin/rctview.asp?TC=1150)
* A history of primary hyperparathyroidism
* A history of osteoporosis for which calcium and Vitamin D treatment are mandatory
* A history of another granulomatous diseases (sarcoidosis, tuberculosis)
* Pregnant or breastfeeding (at index date) female patients
* Patients undergoing other resections than ileocolonic resections
* Patients who prefer to use open-label vitamin D preparations
* Patients who will continue to use tanning beds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with clinically significant endoscopic recurrence at 6 months of vitamin D3 treatment postoperatively, defined as endoscopic Rutgeerts' score ≥i2. | 0-6 months

SECONDARY OUTCOMES:
1. Clinical CD recurrence measured with CDAI among the 2 groups at week 26 (CDAI ≥220) | 0-6 months
2. NOD2 gene mutations: the difference in response to vitamin D treatment in patients NOD2+ versus patients NOD2-. | 0-6 months
3. Difference in significant recurrence among all patients with low vitamin D at baseline | 0-6 months
4. Quality of life, measured by one validated questionnaire for IBD patients (IBD-Q) and two general questionnaires (SF-36 and EuroQol) | 0-6 months
5. Any adverse events | 0-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Geert D'Haens, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Derived] de Bruyn JR, Bossuyt P, Ferrante M, West RL, Dijkstra G, Witteman BJ, Wildenberg M, Hoentjen F, Franchimont D, Clasquin E, van der Bilt JD, Tollens T, Bemelman WA, D'Hoore A, Duijvestein M, D'Haens GR; Dutch-Belgian The Effect of Vitamin D3 to Prevent Postoperative Relapse of Crohn's Disease: A Placebo-controlled Randomized Trial Study Group. High-Dose Vitamin D Does Not Prevent Postoperative Recurrence of Crohn's Disease in a Randomized Placebo-Controlled Trial. Clin Gastroenterol Hepatol. 2021 Aug;19(8):1573-1582.e5. doi: 10.1016/j.cgh.2020.05.037. Epub 2020 May 24. PMID 32461138